CLINICAL TRIAL: NCT05872139
Title: Influence of Exercise/Cardiorespiratory Fitness on Enhanced Endothelial Function With Aging: Role of Mitochondrial-derived Oxidative Stress
Brief Title: Role of Mitochondrial-derived Oxidative Stress to Promote Vascular Endothelial Dysfunction in Non-exercisers With Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Principal Investigator, Brad Fleenor, Associate Professor, Ball State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MitoQ
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Aging; Endothelial Dysfunction; Cardiovascular Function; Arterial Stiffness
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Gelatin capsules
  Interventions: Dietary Supplement: Placebo
- MitoQ (Experimental): Capsules containing mitoquinone mesylate (MitoQ, 5 mg/capsule) totaling 80 mg were taken once.
  Interventions: Dietary Supplement: Mitoquinone Mesylate

INTERVENTIONS:
Dietary Supplement: Placebo — Gelatin capsules
  Arms: Placebo
Dietary Supplement: Mitoquinone Mesylate — MitoQ was given once (single dose, 80 mg)
  Other Names: MitoQ
  Arms: MitoQ

SUMMARY:
The primary goal of this intervention is to determine the efficacy of acute mitochondrial-specific antioxidants to improve vascular endothelial function in middle-aged and older (≥45 y) adults who do no perform regular aerobic exercise. In a double-blind, randomized, placebo-controlled crossover design participants with receive both MitoQ and placebo arm of the study. Primary endpoints will include vascular endothelial function assessed by brachial artery flow-mediated dilation and cardiac function assessed via pulse wave analysis. Secondary endpoints will include measures of aortic stiffness assessed by carotid-femoral pulse wave velocity and carotid artery stiffness (e.g. β-stiffness) and elasticity (carotid compliance, distensibility, and Youngs elastic modulus) from ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Resting brachial blood pressure <160 mmHg (systolic)/<100 mmHg (diastolic)
* Body mass index ≤ 35 kg/m2
* Nonsmoker
* Women must be postmenopausal defined as cessation of menses ≥ 1 year.

Exclusion Criteria:

* cardiovascular/metabolic medications
* known clinical disease
* absolute contraindications to exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function | Baseline and Post 1 hour
  Brachial artery flow-mediated dilation (% [relative] and mm [absolute])

SECONDARY OUTCOMES:
Change in cardiovascular function | Baseline and Post 1 hour
  Subendocardial viability ratio (%)
Change in Aortic Stiffness | Baseline and Post 1 hour
  Carotid-femoral pulse wave velocity (meters/second)
Change in carotid artery stiffness - beta-stiffness index | Baseline and Post 1 hour
  Carotid artery Beta stiffness index (AU)
Change in carotid artery compliance | Baseline and Post 1 hour
  Carotid artery compliance (mmHg/mm^2)
Change in carotid artery distensibility | Baseline and Post 1 hour
  Carotid artery distensibility (10^-3/kilopascals)
Change in carotid artery Young's elastic modulus | Baseline and Post 1 hour
  Carotid artery Young's elastic modulus (kilopascals, kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Fleenor, PhD, Principal Investigator — Associate Professor
Locations (1):
- Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No